CLINICAL TRIAL: NCT00724802
Title: Oral Glyceryl Triacetate (GTA) in Newborns With Canavan
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Dr. Gheona Alteresco, Shaare Zedek Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: canavangta
Record Dates: First submitted 2008-06-18; First posted 2008-07-30 (Estimated); Last update posted 2011-06-21 (Estimated); Status verified 2011-06

CONDITIONS: Canavan Disease
Keywords: babies with canavan disease
MeSH Terms: conditions — Canavan Disease | interventions — Triacetin

INTERVENTIONS:
Dietary Supplement: GTA (Glyceryl triacetate) — 0.5 gr/kg x2/day syrup two times a day with increasing dose each 3 days till max 5gr /kg each day for 6 months
  Other Names: No other names are available for this drug
Drug: GTA glyceryl triacetate — 0.5 gr/kg twice a day with increase of 0.5 gr/kg every 3 days up to 5 gr/kg

SUMMARY:
Canavan disease is caused by Aspartoacylase deficiency. There is no treatment for the disease, but there is a food additive that includes acetate . We suggest an early treatment with acetate and a neurologic evaluation, including MRI, after 4 months of treatment. In any case the treatment will be stopped at the age of 22 months, when myelinization is ended.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of Canavan disease

Exclusion Criteria:

* Age above 18 months

Max Age: 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1 (Estimated)
Dates: Start 2008-03; Primary Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
brain MRI at the end of the study | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Gheona Alterescu, M.D., Principal Investigator — Shaare Zedek Medical Center
Locations (1):
- Shaare Zedek Medical Center, Jerusalem, Israel

REFERENCES:
- [Derived] Segel R, Anikster Y, Zevin S, Steinberg A, Gahl WA, Fisher D, Staretz-Chacham O, Zimran A, Altarescu G. A safety trial of high dose glyceryl triacetate for Canavan disease. Mol Genet Metab. 2011 Jul;103(3):203-6. doi: 10.1016/j.ymgme.2011.03.012. Epub 2011 Mar 15. PMID 21474353